CLINICAL TRIAL: NCT05831592
Title: Evaluation of the Validity and Reliability of Muscle Ultrasound in the Detection of Undernutrition
Acronym: SAURON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Forcilles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A00581-42
Record Dates: First submitted 2023-03-10; First posted 2023-04-26 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Undernutrition
Keywords: undernutrition; muscle ultrasound; diagnostic
MeSH Terms: conditions — Malnutrition; Disease

STUDY DESIGN:
Intervention Model Description: Prospective interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic accuracy of muscle ultrasound in undernutrition (Other): All included patients will undergo an muscle ultrasound assessment in undernutrition
  Interventions: Diagnostic Test: Muscle ultrasound

INTERVENTIONS:
Diagnostic Test: Muscle ultrasound — Muscle ultrasound assessment (sensitivity, specificity) in undernutrition in patients

SUMMARY:
In France, the prevalence of undernutrition in hospitalized patients varies from 30 to 50%. Undernutrition is strongly associated with a decrease in the patient's functional abilities and an increase in morbidity and mortality and healthcare expenses. In 2019, the Global Leadership Initiative on Malnutrition (GLIM) published an international consensus report on diagnostic criteria for undernutrition. The diagnostic criteria are numerous, and include etiological criteria such as reduced food intake; an inflammatory setting; symptoms such as anorexia, fatigue; phenotypic criteria such as weight loss, body mass index (BMI), fat to lean mass ratio, fluid retention, and muscle function.

Muscle mass is described as a major diagnostic criterion, since it is on the one hand a direct indicator of protein catabolism related to undernutrition, but also a reflection of functional impairment in the patient, as it is directly associated with functional capacities, autonomy and prognosis. Ultrasound is a reproducible method of muscle assessment. It allows the evaluation of muscle thickness or cross-sectional area of a muscle, the reduction of which, a marker of atrophy, is strongly correlated to its loss of strength and to reference measurements. In addition, ultrasound can be used to assess muscle quality, particularly by evaluating the echogenicity of the muscle. The echogenicity increases when the muscle is altered, linked to the presence of fatty infiltrate and fibrous tissue. The use of ultrasound in the evaluation of the patient's nutritional status, as a tool for assessing muscle function, is developing in the ICU and is associated with an increase in the patient's comorbidities. Studies remain limited to a few patient populations, do not report clear cut-off values to define muscle pathological status, and require more precise definition of ultrasound measurement protocols.

The investigators hypothesize that muscle ultrasound is reliable and valid in the evaluation of muscle function during the screening of undernutrition in a population of patients hospitalized in diabetology-obesity, pneumology, oncology and gastro-nutrition, under 70 years old.

DETAILED DESCRIPTION:
1. Rationale 1.1 Epidemiology and morbidity of undernutrition Undernutrition, whether related to disease, poverty, hunger, war or natural disasters, affects more than one billion people worldwide. In France, an empirical estimate suggests a prevalence of undernutrition among hospitalized patients of about 2 million or 30 to 50%. It should be noted that undernutrition is very common in and out of hospital. It is widely accepted that undernutrition can be caused by a deficit in nutrient intake or malabsorption. However, it is now known that the inflammatory state present during illness is associated with undernutrition.

   1.2 International consensus on the definition of undernutrition

   In 2019, the Global Leadership Initiative on Malnutrition (GLIM) published an international consensus report on diagnostic criteria for undernutrition. The diagnostic criteria are numerous, and include etiological criteria such as reduced food intake; an inflammatory context; symptoms such as anorexia, fatigue; phenotypic criteria such as weight loss, body mass index (BMI), fat to lean mass ratio, fluid retention, and muscle function. GLIM has chosen to select the most relevant criteria among the etiological and phenotypic criteria:
   * Etiological criteria: reduced food intake and inflammatory state of the patient;
   * Phenotypic criteria: weight loss, BMI, and reduced muscle mass. The presence of at least one etiological criterion and one phenotypic criterion is mandatory to make the diagnosis of undernutrition.

   Muscle mass is described as a major diagnostic criterion, since it is on the one hand a direct indicator of protein catabolism related to undernutrition, but also a reflection of functional impairment in the patient, as it is directly associated with functional capacities, autonomy and prognosis. Different measurement tools are suggested, such as bioelectrical impedancemetry, ultrasound or magnetic resonance imaging, leaving the choice of tool to the clinicians, depending on experience and local resources. Handgrip measurement is considered a complementary measure.

   GLIM recommends an assessment of the risk of undernutrition, using validated questionnaires such as the NRS (Nutritional Risk Screening) or the MNA-SF (Mini Nutritional Assessment- Short Form). The degree of severity of undernutrition is only assessed on the basis of phenotypic criteria.

   1.3 Roles of professionals in screening for undernutrition

   In general, and more particularly in the Forcilles hospital, dieticians play a major role in detecting undernutrition. They ensure a prospective watch on the patient's admission to the hospital, with the collection of indicators related to BMI and weight loss, in collaboration with the nurses and care assistants. They also carry out a dietary consultation to clarify the above criteria, to evaluate the reduction of intake and absorption, in collaboration with the physician, and the realization of body composition measurements, such as bio-electrical impedancemetry. The evolution of the definition of undernutrition, with an important place in the muscular and functional evaluation of the patient, implies new actors: the physiotherapist and the Adapted Physical Activity Teacher (APAT). Indeed, they have expertise in the evaluation of the patient's muscular function and functional capacities. As part of their diagnostic assessment, the physiotherapist is used to evaluating muscle function by dynamometry, as well as the patient's functional capacities by field tests or the use of scores. The EAPA also participates in the performance of field tests.

   The collaboration between dieticians, physiotherapists, EAPAs, nurses, care assistants and doctors thus makes it possible to meet the need to screen for undernutrition according to this new definition.

   1.4 Assessment of muscle function

   Physical therapists and EAPAs use different tools to assess different aspects of muscle function, such as strength or walking speed in more functional tests.

   Isometric grip strength is strongly correlated with lower extremity muscle strength, and is a pejorative marker of mobility in weakness. It has been observed a linear relationship between grip strength and patient disability as measured by the Katz independence scale. In addition, grip strength has been shown to be a good predictor of the patient's clinical condition. The measurement of grip strength, using a dedicated dynamometer, also has the advantage of being simple and reproducible and has reference values adjusted for sex and BMI.

   Gait speed is another indicator used to assess muscle function. It is associated with lower limb strength and is a predictor of disability and mobility limitation. Usual walking speed is most often measured over a distance of 4 or 6 m and has reference values adjusted for sex and height.

   Dietitians also participate in the evaluation of muscle function by measuring body composition in terms of lean and fat mass. They perform bioelectrical impedancemetry, which allows estimation of body fat and lean mass volumes by measuring the resistance of biological tissues to a low-intensity, high-frequency sinusoidal electric current through electrodes. This measurement method is simple to use, inexpensive, reproducible and feasible in bedridden patients. It also correlates very well with MRI and reference values are obtained in various adult populations.

   1.5 Muscle ultrasound and undernutrition

   Ultrasound is a reproducible method of muscle assessmen. It allows the assessment of muscle thickness or cross-sectional area of a muscle, the reduction of which is a marker of atrophy and is strongly correlated with its loss of strength and reference measurements. In addition, ultrasound can be used to assess muscle quality, particularly by evaluating the echogenicity of the muscle. Echogenicity increases with muscle damage, related to the presence of fatty infiltrate and fibrous tissue. Complementary measurements such as pennation angle, fascicular length or fibrillations allow to complete the description of the muscle state.

   Muscle ultrasonography is becoming increasingly used among the tools for assessing muscle function, especially in sarcopenia found in many pathological situations. Its use in the evaluation of the patient's nutritional status, as a tool for assessing muscle function, is developing in the ICU and is associated with an increase in the patient's comorbidities. Studies remain limited to a few patient populations, do not report clear cut-off values to define muscle pathological status, and require more precise definition of ultrasound measurement protocols.

   1.6 Research hypothesis

   The investigators hypothesize that muscle ultrasound is reliable and valid in the evaluation of muscle function during the screening of undernutrition in a population of hospitalized patients in diabetology-obesity, pneumology, oncology and gastro-nutrition, under 70 years of age.
2. Objective 2.1 Main objective The main objective of this study is to evaluate the reliability and validity of muscle ultrasound in the context of screening for undernutrition in patients hospitalized in short-stay and follow-up care and rehabilitation of diabetology-obesity, pneumology, oncology and gastro-nutrition.

2.2 Secondary objectives

The secondary objectives will be, in patients hospitalized in short stay and follow-up care and rehabilitation of diabetes-obesity, pneumology, oncology and gastro-nutrition:

* Evaluate the correlation of muscle ultrasound with standard measures of muscle function;
* To compare the diagnostic capacity of muscle function assessment tools on undernutrition;

  3. Type of study: This is a prospective, monocentric, interventional cohort study. The research will be conducted in accordance with the protocol. The duration of the recruitment will be 20 months with a follow-up of the patients during their entire hospitalization in the care unit, i.e. approximately 30 days (average length of stay), i.e. a total duration of the study estimated at 21 months. The study will take place at the Forcilles Hospital, in diabetology-obesity, pneumology, oncology and gastro-nutrition units.

  4. Description of the usual care 4.1 Usual course of treatment

Patients admitted to short-stay and follow-up care and rehabilitation for diabetes-obesity, pneumology, oncology and gastro-nutrition benefit from medical, nursing and rehabilitation examinations and care. All of this care will not be modified within the framework of this protocol. Physiotherapists and dieticians provide their diagnostic assessment and rehabilitation on medical prescription. The EAPAs participate in the functional evaluation of the patient and carry out physical activities adapted to the patient, also on medical prescription.

As part of the screening for undernutrition in our establishment, the dieticians ensure a prospective and systematic collection of the patient's weight and its evolution over the last few months, of his BMI and an evaluation of the food intake, within 48 hours of the patient's admission to the service. The estimation of the patient's intake is done in collaboration with the nursing assistant.

4.2 Nutritional assessment At the patient's admission, a dietetic evaluation is performed by the dietician following the recommendations issued by the French Association of Dieticians-Nutritionists and the HAS. The dietitian collects all the data needed to detect malnutrition, such as weight, height, BMI, albumin level, and grip strength and walking speed (performed by the caregiver and the physiotherapist or the EAPA). The dietician also looks for possible obstacles to feeding such as dental condition, swallowing problems or digestive discomfort The doctor looks for different pathologies impacting digestive absorption such as shortened or shortened stool syndromes, gastrectomies, pancreatic insufficiency etc. He also looks for factors of aggression such as cancers, chronic progressive diseases, infections etc.

All these data allow us to estimate the theoretical nutritional needs of the patient and to adapt the nutritional management. A follow-up of the ingestations is carried out by the dietician in collaboration with the nurses' aides.

4.2.1 Anthropometric measurements When the patient is admitted, the ward's nurses and orderlies measure the patient's weight and height. When the patient can maintain the erect position, a conventional scale and a measuring rod are used for the measurements. If the patient cannot maintain this position, a weighing chair and a laser meter are used.

In order to evaluate the weight loss before hospitalization, the previous weight is sought in a hospitalization report or another recent medical document. A contact with the attending physician is also made in order to obtain information concerning the patient's weight follow-up. When this information is not available, the previous weight given by the patient is collected.

4.2.2 Biological measurements On admission, a biological sample is usually taken from patients at risk of undernutrition in order to measure pre-albumin, albumin and C-reactive protein (CRP).

4.2.3 Measurements of muscle function Measurement of grip strength ("Handgrip") The gripping force is evaluated with the Jamar® hydraulic force gauge by the caregiver. Measurement of the walking speed ("Gait speed")

Walking speed (m/s) is measured on a 4-meter course, in a corridor, by the EAPA or the physiotherapist.

5. Assessment procedure added by the research : Mini-Nutritional Assessment Short Version (MNA-SF) score, Bioelectrical impedancemetry and muscle ultrasound.

6 Statistical aspects

6.1 Calculation of the number of subjects needed

Reproducibility of ultrasound With an expected intraclass correlation coefficient of at least ρ1 = 0.8, a minimum value ρ0 = 0.70 considered acceptable, a number of observations k= 2, a risk α= 0.05, and a power of 80%, it is necessary to include 118 patients for the study of intra- and inter-examiner reproducibility of ultrasound.

Ultrasound Validity:

With an expected sensitivity and specificity of at least 90% and 85%, respectively, an estimated prevalence of muscle impairment of 45% to 60% in our hospitalized patients, for a risk α= 0.05 and a maximum width of the confidence interval of 10%, it is necessary to include between 87 and 109 patients.

Therefore, it will be necessary to include 118 patients to meet the primary objective of evaluating the validity and reliability of peripheral muscle ultrasound.

6.2 General aspects

Descriptive statistics will be based on means (+/- standard deviation) or medians [interquartile range] depending on the distribution of quantitative variables. Qualitative variables will be described in terms of numbers and percentages. Univariate comparisons will use the usual statistical tests after verification of the distribution of the variables (Chi2 or Fisher's test, t-test, anova or their non-parametric equivalents Wilcoxon and Kruskal-Wallis tests). Paired sample tests will be used if necessary.

Tests will be performed at the 5% significance level. The 95% confidence intervals will be provided for each estimate.

The calculations will be done using SPSS v21 IBM and R software (version 3.6.1, http://www.R- project.org ).

6.3 Morbidity and mortality criteria

6.3.1 Length of hospitalization The length of stay is defined as the number of days of presence in the inclusion service, from the patient's admission to the final discharge. Temporary transfers to another hospital department for an examination or an intervention are not considered discharges.

A special statistical treatment will be carried out on the length of hospital stay, given the impact of death on the length of stay.

6.3.2 Mortality Number of deaths out of the total number of patients included. A specific statistical treatment will be performed on the mortality rate.

6.3.3 Katz Activities Daily Living (ADL) Score The Katz ADL score is completed within 48 hours prior to (scheduled) hospital discharge by the patient's caregiver or nurse. The total score is out of 6. A score of less than 3 indicates major dependence, a score of 0 indicates total dependence.

The Katz ADL score will be treated as a discrete numerical variable.

6.4 Analysis of the main objective

Inter- and intra-examiner reliability will be assessed by calculating intra-class correlation coefficients.

Validity will be assessed by calculating the areas under the ROC curve (Receiver Operating Characteristics) and calculating sensitivities, specificities, positive and negative predictive values.

The reference test for the diagnosis of impaired muscle function is bioelectrical impedance. The cut-off values used for the diagnosis of impaired muscle function are those recommended by GLIM : Appendicular Skeletal Muscle Index (ASMI) < 7 kg/M2 in men and < 5.7 kg/m2 in women.

6.5 Secondary objectives

6.5.1 Correlation of muscle ultrasound with standard measures of muscle function Measures of association between quantitative variables will be performed using Pearson's or Spearman's correlation coefficients depending on the distribution of the data. Measures of association between qualitative variables will be performed using the Chi-square or Fisher test depending on the distribution of the data.

The agreement between quantitative variables will be evaluated using the Bland-Altman method and that between qualitative variables using the Kappa coefficient.

6.5.2 Compare the diagnostic capacity of muscle function assessment tools on undernutrition The diagnostic capabilities of the different tools for measuring muscle function (Handgrip, gait speed, bioelectrical impedance and muscle ultrasound) will be compared by ROC curves.

6.5.3 Evaluate the association of muscle ultrasound measurements with patient morbidity and mortality Morbidity and mortality will be compared between the groups with and without ultrasound-determined muscle function impairment, comparing length of hospital stay, mortality, and independence at discharge.

Length of hospitalization There is a relationship between the incidence of mortality and all of the length of stay variables. Length of stay will therefore be analyzed using a competitive risk method, which takes into account the fact that patients who die are no longer eligible for length of stay analysis.

The estimator also provides the probability of in-hospital death, so the probability of hospital discharge versus death at any time after study inclusion can be assessed simultaneously.

Mortality rate The estimation of mortality rates will be performed by the Kaplan and Meier method. Comparison of the 2 curves will be performed by a Logrank test. The mortality rates in the 2 groups will be estimated via the survival curves.

ADL The ADL score will be compared between the 2 groups using the discrete numerical variable comparison tests described in the general aspects.

7. Expected results in terms of scientific and professional advances The results of this study will make it possible to verify whether ultrasound is a reliable and valid tool in the evaluation of peripheral muscle function in the context of screening for undernutrition. On the other hand, they will allow us to propose threshold values for the alteration of muscle function and to provide information on the ultrasound characteristics of the muscle in the undernourished patient and their association with the prognosis of the patient. The different tools could lead to a different estimation of the reduction of muscle mass and therefore a different prevalence of undernutrition. The results of our study will help to evaluate this and to guide professionals in the choice of tools to assess muscle function.

8 Expected benefits and risks for patients 8.1 Minimal risks and constraints added by the research

All medical and paramedical examinations and management are usually performed except for the MNA-SF questionnaire, muscle ultrasound and bioelectrical impedancemetry, which will be performed systematically in the patients included. The MNA-SF questionnaire is very quick (less than 5 minutes) and therefore causes very little inconvenience to the patient apart from an additional visit by a caregiver. Bioelectrical impedancemetry is a tool for assessing body composition using electrodes applied to the skin surface. The examination lasts an average of 15 minutes and is non-invasive and painless. The minimal constraint is related to the placement of the electrode and the duration of the examination. The ultrasound is also non-invasive and painless. The 3 ultrasounds performed will last about 30m. The minimal constraint is related to the installation of the ultrasound probe and the duration of the examination.

8.2 Expected benefits for the patient

Ultrasound is a relatively simple and inexpensive tool compared to other methods of measuring body composition (DEXA or MRI) and provides additional information on muscle quantity and quality compared to the usual tools for measuring muscle function (Handgrip, functional tests). The results of this study will make it possible to propose to the patient a reliable and valid evaluation tool, more easily available and less restrictive in the evaluation of the muscular quality during undernutrition. This could lead to a wider and more precise evaluation of this muscular impairment in order to propose more adapted therapeutic solutions (exercise training, weight training, nutrition).

ELIGIBILITY:
Inclusion Criteria:

* Admitted in short stay and follow-up care and rehabilitation of diabetology-obesity, pneumology, oncology and gastro-nutrition;
* Age between 18 and 70 years at inclusion;
* Affiliation with a social security system or beneficiary of such a system ;
* Oral, free, informed and express consent of the patient or his/her family member.

Exclusion Criteria:

* Impossible to perform the ultrasound;
* Impossibility of performing bioelectrical impedancemetry ;
* Incapacity to consent;
* Patient refusal to participate in the study;
* Pregnancy (a pregnancy test should be performed if in doubt);
* Breastfeeding woman;
* Person subject to a safeguard of justice measure ;
* Patient under guardianship or curatorship;
* Patient in care limitation;
* Sampling in the ineligible study group.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Reduction in muscle mass measured by ultrasound thickness of the rectus femoris. | Through study completion, an average of 2 years
  The primary endpoint is the reduction in muscle mass measured by ultrasound thickness of the rectus femoris. The reduction in muscle mass measured by ultrasound will be used to estimate the diagnostic accuracy of muscle ultrasound using bioelectrical impedancemetry as the reference examination.

SECONDARY OUTCOMES:
Correlation measurements of muscle ultrasound with: | Through study completion, an average of 2 years
  * Bioelectrical impedancemetry ;
  * Handgrip (using a dynamometer);
  * Walking speed (walking speed is measured over a distance of 4 or 6 m and has reference values adjusted for sex and height).
Comparison of the diagnostic accuracy in undernutrition of muscle ultrasound with those of : | Through study completion, an average of 2 years
  * Bioelectrical impedancemetry;
  * Handgrip (using a dynamometer);
  * Walking speed (walking speed is measured over a distance of 4 or 6 m and has reference values adjusted for sex and height).
Measure of association of muscle ultrasound measurements with patient morbi- mortality: | Through study completion, an average of 2 years
  * Length of hospitalization (days);
  * Mortality: proportion and date of occurrence of death among patients included during hospitalization;
  * ndependence in Activities of Daily Living score (SCORING: 6 = High (patient independent) 0 = Low (patient very dependent)

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric LE NEINDRE, PhD, Principal Investigator — Hopital Forcilles; Virginie COLELLA, MSc, Study Director — Hopital Forcilles
Locations (1):
- Hôpital Forcilles, Férolles-Attilly, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
The protocole, the statistical analysis plan and data will be available as supplementary materials with the publication. The other data that support the findings of this study will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At publication for 10 years
Access Criteria: The data that support the findings of this study will be available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats AJS, Crivelli AN, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee, GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. J Cachexia Sarcopenia Muscle. 2019 Feb;10(1):207-217. doi: 10.1002/jcsm.12383. PMID 30920778
- [Background] Correia MI, Waitzberg DL. The impact of malnutrition on morbidity, mortality, length of hospital stay and costs evaluated through a multivariate model analysis. Clin Nutr. 2003 Jun;22(3):235-9. doi: 10.1016/s0261-5614(02)00215-7. PMID 12765661
- [Background] Biolo G, Cederholm T, Muscaritoli M. Muscle contractile and metabolic dysfunction is a common feature of sarcopenia of aging and chronic diseases: from sarcopenic obesity to cachexia. Clin Nutr. 2014 Oct;33(5):737-48. doi: 10.1016/j.clnu.2014.03.007. Epub 2014 Mar 29. PMID 24785098
- [Background] Nijholt W, Scafoglieri A, Jager-Wittenaar H, Hobbelen JSM, van der Schans CP. The reliability and validity of ultrasound to quantify muscles in older adults: a systematic review. J Cachexia Sarcopenia Muscle. 2017 Oct;8(5):702-712. doi: 10.1002/jcsm.12210. Epub 2017 Jul 12. PMID 28703496

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT05831592/Prot_SAP_ICF_000.pdf